CLINICAL TRIAL: NCT05232305
Title: Evaluation of the Effect of Pomegranate Peel on Plasma Glucose, Lipid Parameters, and Lipid Oxidation in Individuals With Type 2 Diabetes: A Randomized Controlled Study
Brief Title: Evaluation of the Effect of Pomegranate Peel Added Bread on Blood Sugar, Fats, and the Body's Defense Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Toros University (Other)
Responsible Party: Principal Investigator, Özlem ÖZPAK AKKUŞ, Principal Investigator, Toros University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pomegranatepeelintype2DM
Record Dates: First submitted 2021-12-09; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes
Keywords: Antioxidant; Obesity; Pomegranate peel; Oxidation; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Intervention Model Description: The study will conduct by using a prospective randomized double-blind clinical trial model.
Who Masked: Participant, Care Provider
Masking Description: Participants will not know which type of bread to eat.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People with type 2 diabetes who eat bread with pomegranate crust - Experimental Group (Experimental): Individuals with type 2 diabetes who met the inclusion criteria and participated in the study will divided into two groups by Specialist Akkız Zuhal ÖZTAŞ and Specialist Doctor Emel ŞENOL, and they will be asked to consume the breads produced (in the preliminary study) produced as a standard (n=15) and with the addition of pomegranate peel (n=15) for eight weeks.
  The individuals participating in the study will be asked not to change their eating habits, physical activity habits, and drug treatments during the study period. Each individual participating in the study will be provided with the required amount of bread during the study and will be contacted weekly by Zeynep ÇAMLIK, a specialist dietitian, to verify whether they consume bread regularly.
  Interventions: Dietary Supplement: Pomegranate Peel
- No intervention - Control Group (No Intervention): Individuals with type 2 diabetes will not eat pomegranate crust bread

INTERVENTIONS:
Dietary Supplement: Pomegranate Peel — Standard bread and test breads (with added pomegranate peel) to be used in the study will be produced by Asst. Prof. Özlem ÖZPAK AKKUŞ in the Nutrition Principles Laboratory of Toros University. For standard bread, 900 ml of water, 42 fresh yeast, 12 g of salt and 12 g of sunflower oil will be added to 1000 g of sifted whole wheat flour and the prepared bread mixture will be divided into 40 equal parts. To make bread with pomegranate peel added, 1000 g of sifted whole wheat flour, 20 g of pomegranate peel powder, 914 ml of water, 42 g of fresh yeast, 12 g of salt and 12 g of sunflower oil will be added and the prepared bread mixture is divided into 40 equal parts with 500 mg of pomegranate peel powder in each piece).
  Arms: People with type 2 diabetes who eat bread with pomegranate crust - Experimental Group

SUMMARY:
The aim of this study is to evaluate the effects of the consumption of bread produced with the addition of pomegranate peels, which has a high antioxidant content, on blood glucose and lipid parameters, and some oxidant-antioxidant enzymes and lipid peroxidation in individuals with type 2 diabetes.

DETAILED DESCRIPTION:
Between 01.02.2022 and 30.05.2022 with Specialist Dr. Emel SENOL's approval, by Specialist Dr. Akkız Zuhal ÖZTAŞ

The study will be conducted with 30 volunteers who present to the City Hospital Internal Medicine Polyclinic in Mersin.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with type 2 diabetes for at least 5 years,
* Using only oral antidiabetic
* With a Body Mass Index (BMI) value ≥ 25.0 kg/m2,
* Signing the Informed Voluntary Consent Form,
* Being in an age range of 19-64 years.

Exclusion Criteria:

* Having kidney, liver, and inflammatory diseases,
* Being on insulin therapy,
* Using prescription drugs and/or fiber supplements,
* Taking vitamin and mineral supplements,
* Being pregnant/lactating,
* Consuming excessive alcohol (>2 drinks/day),
* Being in the menstrual period,
* Receiving gluten enteropathy,
* Having allergy against pomegranate.
* In addition, individuals with Covid-19-related condition during the study process will be excluded from the study.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Biochemical Blood Parameters | First day at the beginning of the study
  Examination of between group differences regarding lipid profile
Biochemical Blood Parameters | First day at the beginning of the study
  Examination of between group differences regarding HbA1c
Biochemical Blood Parameters | First day at the beginning of the study
  Examination of between group differences regarding insulin
Biochemical Blood Parameters | First day at the beginning of the study
  Examination of between group differences regarding TAC
Biochemical Blood Parameters | First day at the beginning of the study
  Examination of between group differences regarding TBARS
Anthropometric Measurements - Weight | First day at the beginning of the study
  Examination of between group differences regarding weight in kilogram
Anthropometric Measurements - Height | First day at the beginning of the study
  Examination of between group differences regarding height in meter
Anthropometric Measurements - Body Mass Index | First day at the beginning of the study
  Examination of between group differences regarding body mass index (BMI = weight in kilogram / height in meter 2)
Anthropometric Measurements - Waist Circumference | First day at the beginning of the study
  Examination of between group differences regarding waist circumference in centimeters
Anthropometric Measurements - Hip Circumference | First day at the beginning of the study
  Examination of between group differences regarding hip circumference in centimeters

SECONDARY OUTCOMES:
Biochemical Blood Parameters | Eight weeks after the start of the study
  Comparison of between group differences regarding lipid profile
Biochemical Blood Parameters | Eight weeks after the start of the study
  Comparison of between group differences regarding HbA1c
Biochemical Blood Parameters | Eight weeks after the start of the study
  Comparison of between group differences regarding insulin
Biochemical Blood Parameters | Eight weeks after the start of the study
  Comparison of between group differences regarding TAC
Biochemical Blood Parameters | Eight weeks after the start of the study
  Comparison of between group differences regarding TBARS
Anthropometric Measurements - Weight | Eight weeks after the start of the study
  Examination of between group differences regarding weight in kilogram
Anthropometric Measurements - Height | Eight weeks after the start of the study
  Examination of between group differences regarding height in meter
Anthropometric Measurements - Body Mass Index | Eight weeks after the start of the study
  Examination of between group differences regarding body mass index (BMI = weight in kilogram / height in meter 2)
Anthropometric Measurements - Waist Circumference | Eight weeks after the start of the study
  Examination of between group differences regarding waist circumference in centimeters
Anthropometric Measurements - Hip Circumference | Eight weeks after the start of the study
  Examination of between group differences regarding hip circumference in centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Özlem ÖZPAK AKKUŞ, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared in consultation with the principal investigator.
Time Frame: data can be shared after the research is published in consultation with the principal investigator.
Access Criteria: data can be shared after the research is published in consultation with the principal investigator.